CLINICAL TRIAL: NCT01136603
Title: Abdominal Wall Closure After TRAM / DIEP Flap - Comparison of TIGR Mesh vs Polypropylene Mesh.
Brief Title: TIGR vs Polypropylene (Permanent) Mesh: Randomised Trial
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: LIM THIAM CHYE / Professor, National University Hospital / National Unviersity of Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NUHS/SUR-PRAS/2010/2; D / 10 / 344 (Registry Identifier: DSRB: D/ 10 / 344)
Record Dates: First submitted 2010-06-02; First posted 2010-06-03 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Hernia
Keywords: Abdominal wall defects; Inflammation reactions; Amount of tissue ingrowth; Adhesion formation; Shrinkage profiles of the implant
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TIGR Mesh (Experimental): Experimental - TIGR Mesh
  Interventions: Device: TIGR Mesh
- Control (Active Comparator): Control group - Non absorbable Polypropylene mesh
  Interventions: Device: TIGR Mesh

INTERVENTIONS:
Device: TIGR Mesh — TIGR mesh as a reconstruction material for the repair of the abdominal wall post Lipectomy, TRAM / DIEP flap.
  Other Names: Experimental - TIGR Matrix Surgical Mesh; Control - Polypropylene mesh

SUMMARY:
Hypothesis: TIGR mesh as a reconstruction material is a more effective mesh for the repair of the abdominal wall post lipectomy, transverse rectus abdominis myocutaneous (TRAM) / deep inferior epigastric perforator (DIEP) flap.

DETAILED DESCRIPTION:
In this study we will be conducting a randomized trial to study the efficacy of TIGR as a preferred reconstruction mesh for the repair of the abdominal wall post lipectomy, TRAM / DIEP flap.

Aims -

1. Investigating the efficacy of TIGR as a preferred reconstruction mesh for the repair of the abdominal wall post lipectomy, TRAM / DIEP flap. Efficacy of TIGR will allow us to determine the stability of the material in the abdominal wall reconstruction.
2. Study the absorption characteristics of TIGR implant as compared with a non absorbable polypropylene mesh. Absorption characteristics can be determined by the amount of tissue ingrowth, adhesion formation and shrinkage profiles of the implant and it can be detect using ultrasound.
3. To determine whether any reactions to the implant will occur. These reaction if any will manifest as inflammation reactions which may be evident on clinical followup and can be detect by ultrasound.

Patients to be recruited :

80 randomized equally into the 2 groups Age range: 21 - 80 All patients undergoing lipectomy, TRAM / DIEP flap reconstruction will be recruited into the study.

Trial Duration: July 2010 - July 2015

Follow up:

Postoperative 1 week, 1 month, 3 months, 6 months, and 12 months Ultrasound will be done to determine the amount of tissue ingrowth, adhesion formation and shrinkage profiles of the implant in all these follow up appointments. Complications if any can also be detected by the Ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 - 80 years
* Both Male, Female
* all patients undergoing Lipectomy, TRAM / DIEP flap reconstruction
* patients with abdominal wall defects

Exclusion Criteria:

* patient refusal
* infection of the abdominal / generalised infection

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-07; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Shrinkage profiles of the implant | 1 year
  Assess the shrinkage profiles of the implant after implantation using Ultrasound at 1 week, 1 month, 3 months, 6 months and 12 months

SECONDARY OUTCOMES:
Amount of tissue ingrowth | 1 year
  Assess the amount of tissue ingrowth after implantation using Ultrasound at 1 week, 1 month, 3 months, 6 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Thiam Chye Lim, MD, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore, Singapore